CLINICAL TRIAL: NCT00982969
Title: The Clinical Utility of QuantiFERON in the Diagnosis of Active Tuberculosis Among Young Adults
Brief Title: The Clinical Utility of QuantiFERON in the Diagnosis of Active Tuberculosis
Status: Completed | Type: Observational
Sponsor: Armed Forces Capital Hospital, Republic of Korea (Other Government)
Responsible Party: Sei Won Lee/Division chief of pulmonology, Armed Forces Capital Hospital
Other Study IDs: QFTinROKmilitary
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2009-09

CONDITIONS: Tuberculosis
Keywords: tuberculosis; pneumonia; QuantiFERON-TB Gold in-tube; Tuberculin skin test
MeSH Terms: conditions — Tuberculosis; Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TB suspected: Soldiers who are clinically suspected with tuberculosis

SUMMARY:
The investigators will evaluate the usefulness of QuantiFERON-TB Gold in-tube (QFT) in the diagnosis of active tuberculosis in young adults group, highly clinically suspected tuberculosis.

DETAILED DESCRIPTION:
Investigators will enroll prospectively all clinically and radiologically suspected tuberculosis patients from 20 to 29 years old who visited the Armed Forces Capital Hospital. Investigators will perform QFT and tuberculin skin test. Diagnosis of tuberculosis will be made by World Health Organization guideline and the physician will not know the QuantiFERON-TB Gold in-tube results before the diagnosis and anti-tuberculosis medication. Investigators will evaluate the sensitivity and specificity of QuantiFERON-TB Gold in-tube in the diagnosis of active tuberculosis among young adults.

ELIGIBILITY:
Inclusion Criteria:

* All clinically and radiologically suspected TB patients from 20 to 29 years old who visited the Armed Forces Capital Hospital

Exclusion Criteria:

* Soldiers who do not agree with study protocol

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Soldiers in South Korean Army
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Capital Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lee JE, Kim HJ, Lee SW. The clinical utility of tuberculin skin test and interferon-gamma release assay in the diagnosis of active tuberculosis among young adults: a prospective observational study. BMC Infect Dis. 2011 Apr 18;11:96. doi: 10.1186/1471-2334-11-96. PMID 21501477